CLINICAL TRIAL: NCT06029686
Title: Vibrotactile Coordinated Reset for Parkinson's Patients of a More Variable Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vivek P. Buch, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71725
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stimulation (Experimental): Patients will be asked to stimulate using a non invasive vibrotactile device.
  Interventions: Device: Stanford Glove

INTERVENTIONS:
Device: Stanford Glove — The vibrotactile device sends weak non-painful pattern type vibratory stimulus to the fingertips and is non-invasive. Some patient may experience dyskinesia which can me medicated with a decrease in Parkinson's medication

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on Parkinson's symptoms of a more variable population. vCR will be administered with a device called the Stanford Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as Levodopa and or deep brain stimulation. Patients will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 35 - 92 years
2. Idiopathic Parkinson's Symptoms between Hoehn and Yahr stages 2 to
3. Fluent in English
4. Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
5. Feels comfortable going off PD related medication during in person study visits
6. Lives in the United States

Exclusion Criteria:

1. Any significant neuro-psychiatric problems, including acute confusional state, ongoing psychosis, or suicidal tendencies
2. Any current drug or alcohol abuse.
3. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
4. Pregnancy, breast-feeding or wanting to become pregnant
5. Craniotomy
6. Brain surgery
7. Patient is unable to communicate properly with staff (i.e., severe speech problems)
8. Excessive drooling
9. Patient is taking a medication that may cause significant withdrawal effects

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Parkinsonian symptoms as defined by the change in Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III Score | 6 months
  Change in MDS-Unified Parkinson's Disease Rating Scale Part III Scale Score Mean change in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score.
  Minimum score - 0 indicates normal functioning Maximum score - 132 indicated severe impairment
  Lower scores indicate greater functionality and higher scores indicate severe impairment in functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Tass, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No